CLINICAL TRIAL: NCT07092280
Title: A Pilot Study of Transcranial Direct Current Stimulation (tDCS) in Children With Autism Spectrum Disorder
Brief Title: Transcranial Direct Current Stimulation in Children With Autism
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Institute for Basic Research (Other Government)
Responsible Party: Principal Investigator, Helen Yoo, Research Scientist; Head of Applied Behavior Analysis Laboratory, New York State Institute for Basic Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NKI2024-46-IBRDD
Record Dates: First submitted 2025-07-17; First posted 2025-07-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Executive Dysfunction
Keywords: transcranial direct current stimulation; applied behavior analysis
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: sham vs. active transcranial direct current stimulation (tDCS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Active stimulation first, then crossover to Sham stimulation. Each participant will receive BOTH sham and active tDCS but the order of each will be randomized. The active tDCS and sham are procedurally identical. Participants in both arms will have the initial tingling sensation and the active tDCS stimulation will CONTINUE for 20 minutes at 1 mA (milliamps). All tDCS sessions will occur during ABA therapy.
  Interventions: Device: Active tDCS
- Sham tDCS (Sham Comparator): Sham stimulation first, then crossover to Active stimulation. Each participant will receive BOTH sham and active tDCS but the order of each will be randomized. The active tDCS and sham are procedurally identical. Participants in both arms will have the initial tingling sensation, except in sham stimulation, the current will be DISCONTINUED after 30 seconds while the power indicator remains on for the remainder of 20 minutes at 0 mA (milliamps). All tDCS sessions will occur during ABA therapy.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Active tDCS — Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method used to modulate cortical excitability, which produces facilitatory or inhibitory effects on behaviors. The anodal electrode will be positioned at F3 (using the international 10-20 EEG system) to target the left dorsolateral prefrontal cortex (DLPFC). The cathodal electrode will be placed over the right DLPFC. Participants will undergo 20 active stimulation sessions, each lasting 20 minutes at a continuous 1.0 mA intensity.
  Arms: Active tDCS
Device: Sham (No Treatment) — The anodal electrode will be positioned at F3 (according to the international 10-20 EEG system), targeting the left dorsolateral prefrontal cortex (DLPFC). The cathodal electrode will be placed over the right DLPFC. Participants will receive 20 sessions of sham stimulation, each 20 minutes long. At the start of each session, the current ramps up and remains active for 30 seconds. After 30 seconds, the current is DISCONTINUED (held at 0 mA) but the power indicator stays illuminated for the remainder of the 20-minute session to ensure effective blinding, as is standard in tDCS sham protocols
  Arms: Sham tDCS

SUMMARY:
Although many children diagnosed with autism spectrum disorder (ASD) make significant progress in learning and their cognitive skills improve with applied behavior analysis (ABA), there are a significant number of children who show an absence or a plateau in various skills. Deficits in executive functioning are likely to be involved in many of these cognitive and learning disabilities due to poor functioning of the prefrontal cortex. Currently, the use of biological methods for improving learning and cognition is largely unexplored in research and practice.

The aim of this study is to use of transcranial direct current stimulation (tDCS) in combination with ABA to improve the acquisition of educational programs for students with ASD. tDCS is a low-level electrical neurostimulation and is most effective when used in combination with an active training or teaching, facilitating the neuronal circuits used for that task.

tDCS has been used for various indications over a couple of decades and has been shown to be very safe and has been well-tolerated by children with ASD. The mechanism of tDCS is not clear, however animal studies show that tDCS can stimulate the flow of calcium ions through channels in the astrocytes, activating them, and facilitating their role in synapse formation and therefore learning.

DETAILED DESCRIPTION:
Children with ASD experience a wide range of outcomes, and not all children respond effectively to behavioral interventions. This study uses a novel biologic intervention that combines electrical brain stimulation with ABA treatment to target some of the cognitive deficits in ASD that until now have been relatively refractory to treatment.

There is accumulating evidence of tDCS being effective in treating the comorbidities as well as the core symptoms of ASD. tDCS is most effective when used simultaneously with an active intervention. In this study, the effects of tDCS alone and in combination with ABA on the executive functioning skills and the core symptoms of ASD will be examined and monitored using an objective neurophysiological test (EEG).

This is a double-blind, sham-controlled crossover study involving 20 participants. tDCS will be administered while ABA therapy is being implemented. Programs aimed at language and other cognitive functions will be emphasized. tDCS will be applied bi-frontally with the anode at F3 and the cathode at F4. Forty stimulation sessions will be done (20 active, 20 sham) lasting 20 minutes per session, at 1 milliampere.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 5 and 12 years with autism
2. Enrolled in an ABA program (school or in-home) supervised by a Board Certified Behavior Analyst (BCBA)
3. Stable medical and behavioral treatments for at least 4 weeks prior to, and during the study
4. Able to tolerate wearing tDCS as determined during a week-long daily desensitization training.

Exclusion Criteria:

1. Any implanted metal device (heart pacemaker, cochlear implant, surgical clips, etc.)
2. Severe neurological disorders such as TBI, brain tumor, intracranial infection
3. Seizure disorder with a seizure within the last two years
4. Skull defect
5. Peripheral blindness or deafness
6. Medication that might affect tDCS: There have been a few studies concerning the effect of various medications on tDCS. Some may block and others may enhance the effects depending on many factors. The assay used to test these medications was its effect on the motor cortex after stimulation and this may not apply to our montages, however, in order to minimize the chances of having medication affect our results, participants taking the following medications will be excluded:

   * Na or Ca channel blockers which will include all anti-seizure medications
   * Medications that affect the NMDA receptors including dextromethorphan, cycloserine
   * Serotonin reuptake inhibitors
   * Dopamine stimulating or blocking medications including pergolide, bromocriptine and all antipsychotic medications
   * Norepinephrine stimulating or blocking agents including propranolol and the stimulants
   * Drugs that can lower seizure threshold [imipramine, amitriptyline, doxepin, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, phencyclidine, ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline]
   * Barbiturates, benzodiazepines, meprobamate, chloral hydrate in the past 4 weeks
7. Acute skin disease
8. History of magnetic or electrical stimulation

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Behavior Rating Inventory of Executive Function (BRIEF) | Change measured once per month (at the end of each phase) for 5 months
  The BRIEF is a parent-reported executive function questionnaire which utilizes T-scores, which has a mean of 50 with a standard deviation of 10, with a range of 10-100
Change in Electrodncephalogram (EEG) | Change measured once per month (at the end of each phase) for 5 months
  Power, sample entropy, Lyapunov exponent, detrended fluctuation analysis, correlation dimension, and recurrence quantitative analysis (RQA) values on all frequency bands (delta, theta, alpha, beta, gamma, and gamma+) will be computed from 2-minute resting EEGs using a portable headset

SECONDARY OUTCOMES:
Change in the Pervasive Developmental Disorder Behavior Inventory (PDDBI) | Change measured once per month (at the end of each phase) for 5 months
  The PDDBI is a parent-reported questionnaire about the symptoms of ASD. The PDDBI utilizes T-scores, which has a mean of 50 with a standard deviation of 10, with a range of 10-100. The higher the Approach/Withdrawal Problems and the higher the Autism scores, the more severe the deficits. The higher the Receptive/Expressive Social Communication scores, the better the competence in these areas
Change in discrete trial training (DTT) data from applied behavior analysis (ABA) therapy | Obtained once at the completion of the study (5 months after the start of the study).
  Individualized behavior data from ABA therapy. Individualized treatment data may be measured as: response rate per minute/hour/day, percent accuracy, percent interval, and percent correct.

OTHER OUTCOMES:
Vineland Adaptive Behavior Scales (for demographic purposes) | Once during 4-week baseline for the entire study.
  Parent reported daily living skills. Higher scores indicate better competence. The possible range for these scores is typically from 20 to 160 with a mean of 100 and a standard deviation of 15.
Leiter-3 nonverbal intelligence assessment (for demographic purposes) | Once during 4-week baseline (if a similar test was not done in the past three years) for the entire study.
  Nonverbal intelligence test. Higher scores indicate better competence, with a mean of 100 and a standard deviation of 15. Scores can range from Extremely Low (69 and below) to Very Superior (130+).

CONTACTS AND LOCATIONS:
Overall Officials: J. Helen Yoo, Ph.D., Principal Investigator — New York State Institute for Basic Research
Locations (1):
- New York State Institute for Basic Research, Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact jhelen.yoo@opwdd.ny.gov
Supporting Information: Study Protocol, ICF
Time Frame: Start date: January 2026 End date: December 2029
Access Criteria: Researchers engaging in independent scientific research will be provided IPD via email.